CLINICAL TRIAL: NCT06292754
Title: Augmentation of Rotator Cuff Repair With Biodegradable Magnesium Pin: From Bench Side to Bedside
Brief Title: Rotator Cuff Repair With Magnesium Pin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023.211
Record Dates: First submitted 2024-02-05; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Arthroscopic Rotator Cuff Repair
Keywords: ARCR; Magnesium pin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention groups receives treated using magnesium pin in additional to the suture anchor used routinely in clinical practice.
  Interventions: Procedure: magnesium pin in additional to the suture anchor
- Control group (Active Comparator): The control group receives routine suture anchor for the treatment-as-usual (TAU).
  Interventions: Procedure: routine suture anchor

INTERVENTIONS:
Procedure: magnesium pin in additional to the suture anchor — magnesium pin in additional to the suture anchor used routinely in clinical practice
  Arms: Intervention group
Procedure: routine suture anchor — routine suture anchor for the treatment-as-usual
  Arms: Control group

SUMMARY:
Rotator cuff tears are one of the most common conditions encountered in orthopaedic practice leading to significant shoulder pain and functional deficit. The incidence of rotator cuff tears increases with age and previous trauma. Arthroscopic rotator cuff repair (ARCR) is a surgical procedure to reattach the torn edge of the tendon to the underlying bone, which can improve the clinical symptoms of patients. However, the retear rate after arthroscopic repair is as high as 94% (1). The high re-tear rate following cuff repair is due to the lack of a strong tendon to bone integration. The natural healing responses after surgical reattachment are too weak to regenerate strong tendon insertion, primarily owing to insufficient osteogenesis. To enhance the bone-tendon interface (BTI) healing, the investigators have developed a magnesium pin that can be applied to the cuff repair site to improve the BTI healing.This study is a single-center, randomized controlled trial to investigate the effect of using magnesium pin as a suture to augment rotator cuff repair. The intervention groups receives treated using magnesium pin additional to the suture anchor used routinely in clinical practice, whereas the control group receives routine suture anchor for the treatment-as-usual (TAU). The investigators hypothesize the magnesium pin applied in arthroscopic rotator cuff tears can promote BTI healing and reduce the cumulative retear rate with better functional outcomes.

DETAILED DESCRIPTION:
Mechanical enhancement is a direct approach to enhance the bone-tendon interface (BTI) healing, which includes surgical techniques that seek to improve BTI healing through better fixation device. Favourable results would be achieved in the non-massively torn cases, improvement in the structural integrity and shoulder function were reported in the clinical studies. However, despite the improved initial biomechanical strength, high retear rate were still reported among the massive-teared patients, which indicates that enhancing the mechanical enhancement alone may not enough to promote the overall healing outcome. Other novel adjuvants to aid rotator cuff healing to promote bone tendon junction healing include growth factor supplementation, stem cells or biophysical intervention (5,6,7).

Tissue engineering is a promising strategy that would combine modern engineering techniques with novel biomaterials, cell therapy, growth factors, bioactive molecular. Enhancement of BTI healing with biomaterial, such as magnesium, may promote osteogenesis and thus improve the surgical outcome. These various approaches have been investigated in pre-clinical animal models of rotator cuff repair, yet further investigation to translate these into clinical practice is needed (8).

We have developed a magnesium pin that can be applied to the cuff repair site to improve the BTI healing.

The use of biodegradable materials as implants to stimulate healing has been developed in orthopaedics for decades. Our team and others reported that Mg-based interference screw or suture anchors could upregulate the expression of osteogenic and angiogenic factors experimentally, yet further investigation is still required to translate into clinical practice. However, the potential insufficient mechanical strength of Mg-based implants over the degradation period may result in a loss of fixation or failure of repair, which limits its clinical application. Herein, our novel magnesium pin showed good mechanical properties to be used to enhance the suture anchor commonly used for RCT repair in clinical practice. This can incorporate the benefit of an Mg-based component for its degradation and release of osteogenic and angiogenic by-products, but without the risk of compromising the integrity of the RCT repair site or the potentially osteoporotic bone at the repair site.

40 patients with rotator cuff tear scheduled for arthroscopic rotator cuff repair (ARCR) will be recruited from the Li Ka Shing Orthopaedic Specialist clinic at the Prince of Wales Hospital (PWH) Hong Kong.

Oral and written consents will be obtained from individuals who agree to participate in the study.

The recruitment period will last for 12 months and the whole project period is 2 years in total. Basic demographics, MRI assessment and Outcome Measurement Questionnaires will be carried out.

The intervention groups receive treated using magnesium pin in additional to the suture anchor used routinely in clinical practice, whereas the control group receives routine suture anchor for the treatment-as-usual (TAU). Both treatments are conducted in clinical practices that are randomly allocated to either the intervention or the control condition. Participants are therefore randomized as their allocation depends on their practice being an intervention or a control practice.

Assessments including anthropometric measurement, range of motion, shoulder muscle strength assessment, inflammation test and questionnaires will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires Arthroscopic rotator cuff repair (ARCR) and amenable to repair.
* Subject is > 40 years of age (no upper limit);
* Subject provides written informed consent for study participation using an Independent Ethical Committee (IEC) / Institutional Review Board (IRB) approved consent form;
* Subject is willing and able to participate in required follow-up visits and is able to complete study activities.

Exclusion Criteria:

* Subjects who are unable to tolerate magnetic resonance imaging (MRI), due to psychiatric or medical contraindications;
* Subjects with Samilson-Prieto osteoarthritis > 2;
* Subjects with current or prior infection of the ipsilateral shoulder;
* Subjects with known inflammatory arthropathy, history of inflammatory arthropathy, or chronic joint disease;
* Subjects with prior shoulder surgery (not including rotator cuff repair (revision repair subject group only), biceps tenodesis/tenotomy, distal clavicle excision (DCE), ubacromial decompression);
* Subjects with an irreparable or partially reparable rotator cuff tear;
* Subjects with a subscapularis tear requiring repair;
* Subjects requiring a concomitant labral fixation procedure;
* Subjects requiring a concomitant os acromiale fixation procedure
* Subjects with glenohumeral joint instability (multiple dislocations/subluxations);
* Subjects with a subacromial or intra-articular injection within 3 months prior to surgery;
* Subjects with condition(s) that contraindicate or complicate outcomes of ARCR e.g., > Hamada 3 rotator cuff arthropathy on X-ray, Goutallier atrophy > Grade 3, proximal humeral fracture or scapular fracture, avascular necrosis of the humeral head or glenoid, history of immunodeficiency disorders, history of chronic inflammatory disorders, oral or injected steroid use in last 4 weeks;
* Pregnancy or possibility of pregnancy
* Patient's inability to understand written and spoken Chinese, Mandarin or English.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Imaging Examinations | Baseline, post-operative 3 months, 6 months, and 12 months.
  Upper extremity Magnetic resonance imaging (MRI) for study participants will be collected at Baseline, at 3, 6 and 12 months. The Baseline (pre-operative) MRI follows standard of care imaging and will not follow the study MRI Image Acquisition Protocol. The Baseline MRI must occur within 6 months of enrollment into this study. MRI at 3, 6- and 12-months post-surgery will be collected per Image Acquisition Protocol. Total tendon thickness (mm), tendon length (mm), size of retear (anteroposterior /mediolateral), and shape of retear will be recorded.
Cofield classification | Baseline, post-operative 3 months, 6 months, and 12 months.
  The Cofield classification system will be used for all MRI analyses to assess the size of full-thickness tears(FTT) :
  • Small = < 1 cm • Medium = 1-3 cm • Large = 3-5 cm • Massive = > 5 cm
Sugaya Score | Baseline, post-operative 3 months, 6 months, and 12 months.
  The Sugaya score will be used to determine postoperative cuff integrity through magnetic resonance imaging classified into 5 categories: Type I to Type V. Type I indicates sufficient thickness with homogenously low intensity. Type II indicates sufficient thickness with partial high intensity. Type III indicates insufficient thickness without discontinuity. Type IV indicates presence of a minor discontinuity, suggesting a small full-thickness tear. Type V indicates the presence of a major discontinuity, suggesting a medium or large full-thickness tear.
Goutallier Classification | Baseline, post-operative 3 months, 6 months, and 12 months.
  The Goutallier classification will be used to classify the fatty infiltration of the rotator cuff. The Goutallier classification ranges from a grade of 0 indicating a completely normal muscles without any fatty streaks to a grade of 4 which indicates that more fat than muscle is present . Grade 0: Completely normal muscle, without any fatty streaks, Grade 1: Some fatty streaks, Grade 2: Increased fatty infiltration, but more muscle than fat, Grade 3: Equal amounts of fat and muscle, Grade 4: more fat than muscle.

SECONDARY OUTCOMES:
Height measurement | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  Height will be measured and report in meter.
Weight measurement | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  Weight will be measured and report in kg.
BMI measurement | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  Weight and height will be measured and combined to report Body mass index (BMI) in kg/m^2.
Shoulder flexibility (range of motion) | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  The passive range of shoulder flexion, shoulder abduction and shoulder internal and external rotation will be measured by a goniometer with the participant lying supine. Three measurements will be recorded and averaged for analysis.
Shoulder muscle strength | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  The isometric force of shoulder internal and external rotation will be measured using a handheld dynamometer (HOGGAN Health Industries Inc, West Jordan, Utah). The subject will be asked to push against the examiner's resistance for 5 seconds. Three measurements will be recorded and averaged for analysis. The peak force will be normalized with the participant's body weight.
Western Ontario Rotator Cuff (WORC) Index Western Ontario Rotator Cuff (WORC) Index Index | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  The WORC Index is a 21-item questionnaire assessing quality of life, evaluating the change in symptoms and functional ability, specific to rotator cuff tendinopathy; it is often used to compare pre-and postoperative changes in patients with a clinical diagnosis of an impingement syndrome, rotator cuff tendinopathy as well as arthroscopic rotator cuff repairs (ARCR).Raw scores range from 0 to 2100, with a higher score indicating decreased quality of life because of pathological condition of the rotator cuff.
Constant-Murley Score | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  The Constant-Murley Score is a validated assessment of pain and shoulder functionality. The test is divided into four subscales: pain, activities of daily living, strength and range of motion (forward elevation, external rotation, abduction and internal rotation of the shoulder. The subjective findings (severity of pain, activities of daily living and working in different positions) comprise 35 points and the objective (examiner-assessed) measurements (arm range of motion without pain, measurements of exo- and endorotation via reference points and measuring muscle strength) comprise the remaining 65 points, for a total of 100 points.
Visual Analogue Scale (VAS) | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  Pain is assessed on a 100-point scale ranging from 0 to 100, with zero (0) representing no pain and 100 representing the worst pain imaginable.
Adverse events | baseline, post-operative 2 weeks, 3 months, 6 months, and 12 months.
  Any events related to the surgery will be recorded.
C-reactive protein measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  5 ml blood samples will be collected and analysied for C-reactive protein measurement using a commercially available an enzyme-linked immunosorbent assay (ELISA) kit.
Calcium (Ca) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of calcium (Ca) will be taken to monitor potential effect of magnesium pin.
Magnesium (Mg) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of Mg will be taken to monitor potential effect of magnesium pin.
Phosphorous (P) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of phosphorous will be taken to monitor potential effect of magnesium pin.
Creatinine (Cr) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of Cr will be taken to monitor potential effect of magnesium pin.
Urea measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of urea will be taken to monitor potential effect of magnesium pin.
Alanine transaminase (ALT) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of ALT will be taken to monitor potential effect of magnesium pin.
Aspartate aminotransferase (AST) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of AST will be taken to monitor potential effect of magnesium pin.
Total protein (TP) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of TP will be taken to monitor potential effect of magnesium pin.
Albumin (ALB) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of ALB will be taken to monitor potential effect of magnesium pin.
Globulin (GLB) measurement | baseline, day 1 post-operatively, 2 weeks, 3 months and 6 months post-operatively
  The measurements of GLB will be taken to monitor potential effect of magnesium pin.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers